CLINICAL TRIAL: NCT04489680
Title: Educational Impact and Development of a Novel Cleft Palate Surgical Simulator: Improvement in Surgical Trainees' Knowledge and Confidence.
Brief Title: Cleft Palate Surgical Simulator: Improvement in Surgical Trainees' Knowledge and Confidence.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, zavira heinze, Principle Investigator, Guy's and St Thomas' NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Cleft Palate 3D Simulator
Record Dates: First submitted 2020-06-25; First posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Cleft Palate Lip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical Trainees undergoing Cleft Palate Training (Experimental): 26 UK specialty trainees performed a vomerine mucosal flap and intra-velar veloplasty in a one-hour workshop. Pre- and post-simulation questionnaires assessing cleft knowledge and surgical confidence were compared for statistical significance.
  Interventions: Other: Educational

INTERVENTIONS:
Other: Educational — Teaching session

SUMMARY:
Trainees' experience in cleft surgery is limited due to the high-risk nature of the surgery and centralization of cleft care. Simulations allow trainees to learn complex surgical skills whilst ensuring patient safety. Existing cleft surgical simulators are over-simplified or prohibitively expensive. We developed and tested a high-fidelity yet cost-effective simulator for cleft palate repair.

Skeletal elements were obtained through high-resolution scanning of a pathologic specimen, 3D printed and then molded in plastic. Soft tissue components were formed through molding layers of silicone. 26 UK specialty trainees performed a vomerine mucosal flap and intra-velar veloplasty in a one-hour workshop. Pre- and post-simulation questionnaires assessing cleft knowledge and surgical confidence were compared for statistical significance.

DETAILED DESCRIPTION:
Background: Trainees' experience in cleft surgery is limited due to the high-risk nature of the surgery and centralization of cleft care. Simulations allow trainees to learn complex surgical skills whilst ensuring patient safety. Existing cleft surgical simulators are over-simplified or prohibitively expensive. We developed and tested a high-fidelity yet cost-effective simulator for cleft palate repair.

Methods: Skeletal elements were obtained through high-resolution scanning of a pathologic specimen, 3D printed and then molded in plastic. Soft tissue components were formed through molding layers of silicone. 26 UK specialty trainees performed a vomerine mucosal flap and intra-velar veloplasty in a one-hour workshop. Pre- and post-simulation questionnaires assessing cleft knowledge and surgical confidence were compared for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Plastic Surgery Training Residents

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Cleft lip palate surgical knowledge | Day 1
  The knowledge questionnaire was a 10-part questionnaire, developed through consensus between a panel of expert cleft surgeons. Answers were marked by a single assessor according to the agreed marking criteria and participants received a score of 0-10
Cleft lip palate surgical confidence | Day 1
  The confidence questionnaire was a 10-part questionnaire, each scored on a Likert scale of 1-5 that has previously been published and validated for use in cleft palate surgery(Appendix 3).(18) The total score ranged from 10-50, converted by division of 10 to an overall confidence score of 1-5 with 1 being not at all confident to 5 being very confident/at the level of an attending/consultant surgeon

CONTACTS AND LOCATIONS:
Overall Officials: Kezia Echlin, Principal Investigator — Birmingham Children's Hospital
Locations (1):
- Guys and St Thomas Hospital Plastic Surgery, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
On request
Supporting Information: Study Protocol
Time Frame: Anonymous data will be available on request to the authors. Data will be kept for 15 years minimum.
Access Criteria: The request needs to be done by a practicing clinician, able to provide registration proof.